CLINICAL TRIAL: NCT02465606
Title: An Open-Label Study to Evaluate the Safety of Lebrikizumab Compared to Topical Corticosteroids in Adult Patients With Persistent, Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety of Lebrikizumab Compared to Topical Corticosteroids in Adult Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS29735
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — lebrikizumab; Triamcinolone Acetonide

ARMS (2):
- Group 1: Lebrikizumab Dose Level 1 Monotherapy (Experimental): During the 2-week run-in period, participants will receive topical corticosteroid creams to be self-applied two times per day to active skin lesions only. During the 12-week treatment period, lebrikizumab monotherapy will be administered by subcutaneous (SC) injection, but participants assigned to this group will not receive topical corticosteroids. During the 8-week safety follow-up period, all participants will receive topical corticosteroids to be self-applied to active skin lesions as decided by the participant and study investigator.
  Interventions: Drug: Lebrikizumab; Drug: Topical Corticosteroid Creams (Triamcinolone acetonide 0.1% and Hydrocortisone 2.5%)
- Group 2: Topical Corticosteroid Creams Only (Active Comparator): During the 2-week run-in period and during the 12-week treatment period, participants assigned to this group will receive topical corticosteroid creams to be self-applied two times per day to active skin lesions only. During the 8-week safety follow-up period, all participants will receive topical corticosteroids to be self-applied to active skin lesions as decided by the participant and study investigator.
  Interventions: Drug: Topical Corticosteroid Creams (Triamcinolone acetonide 0.1% and Hydrocortisone 2.5%)

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab Dose Level 1 subcutaneous monotherapy was administered SC once every 4 weeks for a total of 3 doses.
  Arms: Group 1: Lebrikizumab Dose Level 1 Monotherapy
Drug: Topical Corticosteroid Creams (Triamcinolone acetonide 0.1% and Hydrocortisone 2.5%) — Triamcinolone acetonide 0.1% cream will be supplied as single 454-g jars to be used on the body. Hydrocortisone 2.5% cream will be supplied as single 28-g tubes to be used on the face and intertriginous areas as indicated.

SUMMARY:
The primary objective for this study is to evaluate the safety of lebrikizumab compared with Topical Corticosteroids (TCS) alone in patients with persistent moderate to severe Atopic Dermatitis (AD) that is inadequately controlled with TCS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years, inclusive, at the start of the run-in period
* AD diagnosed by the Hanifin/Rajka criteria and that has been present for at least 1 year at screening
* Moderate to severe AD as graded by the Rajka/Langeland criteria at screening
* History of inadequate response to a >/= 1 month (within the 3 months prior to the screening visit) treatment regimen of at least daily TCS and regular emollient for treatment of AD
* EASI score >/= 14 at screening
* IGA score >/= 3
* AD involvement of >/= 10% body surface area
* Pruritus Visual Analog Scale score >/= 3

Exclusion Criteria:

* Past and/or current use of any anti-IL-13 or anti-IL-4/IL-13 therapy, including lebrikizumab
* Use of an investigational agent within 4 weeks prior to screening or within 5 half-lives of the investigational agent, whichever is longer
* Evidence of other skin conditions, including, but not limited to, T-cell lymphoma or allergic contact dermatitis
* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Use of any complementary, alternative, or homeopathic medicines including, but not limited to, phytotherapies, traditional or non-traditional herbal medications, essential fatty acids, or acupuncture within 7 days prior to the run-in period or need for such medications during the study
* Evidence of other skin conditions; including, but not limited to, T-cell lymphoma or allergic contact dermatitis
* Evidence of, or ongoing treatment (including topical antibiotics) for active skin infection at screening
* Other recent infections meeting protocol criteria
* Active tuberculosis requiring treatment within the 12 months prior to Visit 1
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* Known immunodeficiency, including HIV infection
* Use of a topical calcineurin inhibitor (TCI) at the time of screening, unless the patient is willing to stop TCI use during the study (including the run-in period) and, in the investigator's opinion, it is safe to do so
* Clinically significant abnormality on screening ECG or laboratory tests
* Known current malignancy or current evaluation for a potential malignancy, including basal or squamous cell carcinoma of the skin or carcinoma in situ
* History of malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | From baseline to week 12

SECONDARY OUTCOMES:
Immunogenicity: Percentage of participants with anti-Lebrikizumab antibodies | From baseline to week 20
Number of participants with disease rebound following discontinuation of study drug | within 20 weeks
Serum lebrikizumab concentration at Week 12 | Week 12
Elimination half-life | Week 4
Number of participants with skin and other organ system infections | From baseline to week 12
Number of participants with injection site reactions | From baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (12):
  - T. Joseph Raoof Md, Inc., Encino, California
  - Allergy and Asthma Relief Experts, Granada Hills, California
  - Allergy and Asthma Associates of Southern California - CRN, Mission Viejo, California
  - Forward Clinical Trials, Tampa, Florida
  - Dermatology Specialists Research, LLC, Louisville, Kentucky
  - Respiratory Medicine Research; Institue of Michigan P.L.C., Ypsilanti, Michigan
  - Sadick Research Group, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Medical Research Center, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Asthma & Allergy Physicians of Rhode Island Clinical Research Institute (AAPRI CRI), Warwick, Rhode Island
  - Center for Clinical Studies, Cypress, Texas
- Canada (7):
  - Dr. Lorne E. Albrecht Inc., Surrey, British Columbia
  - Skin Care Centre, Vancouver, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Guenther Research Inc., London, Ontario
  - The Centre for Clinical Trials Inc., Oakville, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario